CLINICAL TRIAL: NCT04201119
Title: Effect of Oxiris® Membrane on Microcirculation Following Cardiac Surgery Under Cardiopulmonary Bypass: a Pilot Prospective Monocentric Study (Oxicard Study).
Acronym: OXICARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2019_843_0072
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Surgery; Cardiac Event
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Oxiris (Experimental)
  Interventions: Device: Oxiris
- Without Oxiris (No Intervention)

INTERVENTIONS:
Device: Oxiris — Oxiris membrane used on the Prismaflex device (Baxter) dedicated to that type of membrane at blood pump flow of 450 ml min-1
  Arms: With Oxiris

SUMMARY:
Oxiris membrane is an efficient tool for inflammatory cytokines adsorption. Cardiac surgery is followed by an inflammatory state mimicking sepsis. The investigators hypothesized that cytokine adsorption by Oxiris® membrane can attenuate the inflammatory response and thus decrease the microcirculation impairment that followed cardiac surgery.

DETAILED DESCRIPTION:
Oxiris membrane is an efficient tool for inflammatory cytokines adsorption. Cardiac surgery is followed by an inflammatory state mimicking sepsis. The investigators hypothesized that cytokine adsorption by Oxiris® membrane can attenuate the inflammatory response and thus decrease the microcirculation impairment that followed cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 18 years old
* Elective cardiac surgery under CPB with an expected CPB time > 90 minutes (double valve replacement or valve replacement plus coronary arterial bypass graft (CABG))
* Written informed consent from patient or legal surrogates

Exclusion Criteria:

* Missing informed consent.
* Planned CPB hypothermia <32ºC
* Emergency surgery.
* Acute infective endocarditis.
* Immunosuppressive treatment or steroids (prednisone > 0.5 mg/kg/day or equivalent).
* AIDS with a CD4 count of < 200/ μl
* Autoimmune disorder.
* Transplant receptor.
* Advanced Chronic Kidney Disease (CKD 4 or 5).
* Renal replacement therapy (RRT) in the last 90 days.
* Documented intolerance to study device.
* Inclusion in other ongoing study within the last 30 days.
* Pregnancy.
* Coexisting illness with a high probability of death (inferior to 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Improvement in microcirculatory flow measured by sublingual microcirculation device (SDF/OPS) at day 1 following cardiac surgery with Oxiris membrane during CPB time. | Day 1

SECONDARY OUTCOMES:
Improvement in microcirculation flow with Oxiris® membrane during CPB time at 6 hours after cardiac surgery | at 6 hours
Improvement in microcirculation flow with Oxiris® membrane during CPB time at 2 days after cardiac surgery | at 2 days
Decrease of myocardial infarction with Oxiris® membrane | at day 30
  Major cardiovascular and cerebral events (MACCE) are myocardial infarction, stroke, ischemic mesenteric, cardiac arrest, sudden death, acute kidney injury, In-hospital mortality
Decrease of stroke with Oxiris® membrane | at day 30
  Major cardiovascular and cerebral events (MACCE) are myocardial infarction, stroke, ischemic mesenteric, cardiac arrest, sudden death, acute kidney injury, In-hospital mortality
Decrease of ischemic mesenteric with Oxiris® membrane | at day 30
  Major cardiovascular and cerebral events (MACCE) are myocardial infarction, stroke, ischemic mesenteric, cardiac arrest, sudden death, acute kidney injury, In-hospital mortality
Decrease of cardiac arrest with Oxiris® membrane | at day 30
  Major cardiovascular and cerebral events (MACCE) are myocardial infarction, stroke, ischemic mesenteric, cardiac arrest, sudden death, acute kidney injury, In-hospital mortality
Decrease of sudden death with Oxiris® membrane | at day 30
  Major cardiovascular and cerebral events (MACCE) are myocardial infarction, stroke, ischemic mesenteric, cardiac arrest, sudden death, acute kidney injury, In-hospital mortality
Decrease of acute kidney injury with Oxiris® membrane | at day 30
  Major cardiovascular and cerebral events (MACCE) are myocardial infarction, stroke, ischemic mesenteric, cardiac arrest, sudden death, acute kidney injury, In-hospital mortality
Decrease of In-hospital mortality with Oxiris® membrane | 30 days
  Major cardiovascular and cerebral events (MACCE) are myocardial infarction, stroke, ischemic mesenteric, cardiac arrest, sudden death, acute kidney injury, In-hospital mortality
Decrease of cumulative catecholamine use with Oxiris® membrane in the postoperative care period time | day 30
  catecholamine are dobutamine and norepinephrine
Decrease of Requirement for renal replacement therapy events with Oxiris® membrane | 30 days
Sepsis-related Organ Failure Assessment (SOFA) score with Oxiris® membrane | 30 days
  The quick SOFA score (qSOFA) assists health care providers in estimating the risk of morbidity and mortality due to sepsis.
  The score ranges from 0 to 3 points. The presence of 2 or more qSOFA points near the onset of infection was associated with a greater risk of death or prolonged intensive care unit stay.
Simplified Acute Physiology Score (SAPS) II score with Oxiris® membrane | 30 days
  SAPS II was designed to measure the severity of disease for patients admitted to Intensive care units aged 18 or more.
  24 hours after admission to the ICU, the measurement has been completed and resulted in an integer point score between 0 and 163 and a predicted mortality between 0% and 100%. No new score can be calculated during the stay. If a patient is discharged from the ICU and readmitted, a new SAPS II score can be calculated.
  This scoring system is mostly used to:
  describe the morbidity of a patient when comparing the outcome with other patients.
  describe the morbidity of a group of patients when comparing the outcome with another group of patients
decrease of day number in ICU with Oxiris® membrane | 30 days
decrease of hospital stay in days with Oxiris® membrane | 30 days
Decrease of syndecan-1 expression from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Decrease of syndecan-1 expression from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | day 1
Decrease of syndecan-1 expression from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | day 2
Decrease of heparan-sulfate expression from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Decrease of heparan-sulfate expression from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | day 1
Decrease of heparan-sulfate expression from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | day 2
Decrease of hyaluronic acid expression from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Decrease of hyaluronic acid expression from baseline (prior to surgery) versus 1 day after surgery with Oxiris® membrane | day 1
Decrease of hyaluronic acid expression from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | day 2
Variation of inflammatory cytokine concentration from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of inflammatory cytokine concentration from baseline (prior to surgery) versus 1 day after surgery with Oxiris® membrane | one day
Variation of inflammatory cytokine concentration from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | two days
Variation of endothelin concentration from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of endothelin concentration from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
  - Comparison endothelin from baseline and at the end of cardiac surgery, H6, day 1 and day2
Variation of endothelin concentration from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | 2 days
Variation of angiopoietin 1 concentration from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of angiopoietin 1 concentration from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
Variation of angiopoietin 1 concentration from baseline (prior to surgery) versus two days after surgery with Oxiris® membrane | two days
Variation of angiopoietin 2 concentration from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of angiopoietin 2 concentration from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
Variation of angiopoietin 2 concentration from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | 2 days
Variation of Tie2 soluble receptor concentration from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of Tie2 soluble receptor concentration from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
Variation of Tie2 soluble receptor concentration from baseline (prior to surgery) versus two days after surgery with Oxiris® membrane | two days
Variation of VEGF concentration from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of VEGF concentration from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
Variation of VEGF concentration from baseline (prior to surgery) versus two days after surgery with Oxiris® membrane | two days
Variation of myocardial strain from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of myocardial strain from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
Variation of myocardial strain from baseline (prior to surgery) versus two days after surgery with Oxiris® membrane | two days
Variation of diastolic function from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of diastolic function from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
Variation of diastolic function from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | 2 days
Variation of systolic function from baseline (prior to surgery) versus 6 hours after surgery with Oxiris® membrane | 6 hours
Variation of systolic function from baseline (prior to surgery) versus one day after surgery with Oxiris® membrane | one day
Variation of systolic function from baseline (prior to surgery) versus 2 days after surgery with Oxiris® membrane | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abou-Arab O, Huette P, Haye G, Guilbart M, Touati G, Diouf M, Beyls C, Dupont H, Mahjoub Y. Effect of the oXiris membrane on microcirculation after cardiac surgery under cardiopulmonary bypass: study protocol for a randomised controlled trial (OXICARD Study). BMJ Open. 2021 Jul 9;11(7):e044424. doi: 10.1136/bmjopen-2020-044424. PMID 34244250
- [Derived] Nguyen M, Alvarez M, Evezard C, Ibrahima A, Huette P, Mahjoub Y, Pais-De-Barros JP, Bouhemad B, Masson D, Gautier T, Guinot PG, Abou-Arab O. Impaired endotoxin inactivation, rather than gut translocation, is associated with organ injury in cardiac surgery with cardiopulmonary bypass: An ancilliary analysis of a randomised control trial. Eur J Anaesthesiol. 2026 Jan 14. doi: 10.1097/EJA.0000000000002350. Online ahead of print. PMID 41532670